CLINICAL TRIAL: NCT06965049
Title: Multicentric Clinical Pilot Trial Testing the Association Between Antibiotics and Vaginal Probiotics for Patients With Prematured Rupture of Membranes Between 24 and 32 Weeks of Amenorrhea ( PROB-PROM Study)
Brief Title: Vaginal Probiotics During Pregnancy After Premature (24-32 Weeks of Gestation) Preterm Rupture of Membranes
Acronym: PROB-PROM
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre hospitalier de l'Université de Montréal (CHUM) (Other)
Collaborators: Lallemand Health Solutions, Canada (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MP-02-2025-12882
Record Dates: First submitted 2025-04-14; First posted 2025-05-11 (Actual); Last update posted 2025-05-11 (Actual); Status verified 2025-05

CONDITIONS: Pregnancy; Prematurity; PPROM
Keywords: pregnancy; prematurity; PPROM; vaginal probiotics; microbiota
MeSH Terms: conditions — Premature Birth; Preterm Premature Rupture of the Membranes | interventions — Probiotics

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Research pharmacy will be blinded
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Probiotics group (Active Comparator): Probiotics is a mix of probiotic strains.
  Interventions: Other: Probiotic
- Placebo group (Placebo Comparator): Capsule of sugar, same appearance than the probiotic.
  Interventions: Other: Placebo

INTERVENTIONS:
Other: Probiotic — Participant will take 1 intravaginal capsule once a day at bedtime between inclusion in the study until delivery
  Arms: Probiotics group
Other: Placebo — Participant will take 1 intravaginal capsule once a day at bedtime between inclusion in the study until delivery
  Arms: Placebo group

SUMMARY:
The goal of this clinical trial is to evaluate the feasibility of the randomized controlled trial (RCT).

Secondary objectives include comparing the microbiota of preterm babies born after premature rupture of membranes across study groups.

To achieve this, participants will be asked to:

* Use the vaginal study product from the time of membrane rupture until delivery
* Keep a diary documenting their symptoms and treatment adherence
* Provide vaginal secretion samples and stool samples from their baby

DETAILED DESCRIPTION:
Premature rupture of fetal membranes before labor (PPROM) accounts for 30% of preterm births. Since PPROM is strongly associated with ascending vaginal infection, antibiotics are recommended during the latent period (LP) (the interval between rupture and birth). While they prolong the LP and improve neonatal health, they also exacerbate pre-existing vaginal dysbiosis. The addition of vaginal probiotics (VP) helps stabilize the vaginal microbiota (VM) and increase Lactobacillus levels. By enhancing the presence of beneficial bacteria in the vagina, probiotics help restore the balance between beneficial and pathogenic microbes, potentially reducing uterine infection and improving the fetal intestinal microbiota.

Pathophysiological Hypotheses for Improving Neonatal Health

The use of VP may influence neonatal outcomes through three potential mechanisms:

i) Reduction of vaginal dysbiosis: Prolongs pregnancy and mitigates complications related to fetal immaturity (e.g., decreases risk of intraventricular hemorrhage).

ii) Reduction of intrauterine infection/inflammation: Lowers neonatal complications associated with inflammation (e.g., reduces incidence of cystic periventricular leukomalacia).

iii) Improvement of neonatal intestinal microbiota (NIM) through probiotic ingestion: Decreases complications linked to neonatal dysbiosis (e.g., reduces risk of necrotizing enterocolitis [NEC]).

Primary Objectives

* To assess the validity of:

  i) A recruitment rate > 35% ii) A treatment adherence rate > 80% iii) A sample attrition rate < 5%
* To identify barriers and facilitators in different settings for the implementation of the randomized controlled trial (RCT).

Secondary Objectives

* To compare the presence of probiotics in the vaginal microbiota and neonatal stool (meconium and at 7 days of life).
* To measure the effect of probiotics on the evolution of maternal vaginal microbiota and neonatal intestinal microbiota.

Population Pregnant women aged 18 years or older giving birth at one of the eight centers participating in the study in Quebec and Ontario, Canada. Participants will be randomly assigned, in a blinded manner, to either the probiotic or placebo group.

ELIGIBILITY:
Inclusion Criteria:

* women ≥ 18 years of age;
* mono-fetal pregnancy;
* treated for PPROM between 24 and 32 weeks of gestation with latency period between 12 hours and < 7 days in one of the study centers with expectant management;
* speaking and able to read French or English.

Exclusion Criteria:

* Presence of active labor;
* Situation contraindicating expectant management (e.g., infection);
* Significant malformation, chromosomal anomaly, or fetal death;
* Signs of fetal distress;
* Allergy or intolerance to any of the following substances: vitamin C (ascorbic acid), magnesium stearate, maltodextrin, gelatin, yeast, sucrose, trehalose;
* Allergy to soy or lactose;
* Weakened immune system (e.g., AIDS, prolonged corticosteroid treatment, etc.);
* Vaginal probiotics intake 15 days before study inclusion;
* Oral probiotic intake 30 days before study inclusion.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2025-09-01 (Estimated); Primary Completion 2026-03-01 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
Recruitment rate | 7 months
  To assess the feasibility of the study, each local site team will complete a dashboard documenting every individual met and informed about the study. This dashboard will be used to calculate the recruitment rate, using the formula:
  Recruitment rate = (Number of eligible patients - Number of patients who did not consent) / Number of eligible patients Additionally, the dashboard will track reasons for acceptance or refusal.
Feasability dashboard | 7 months
  The attrition rate will be explored to assess feasability of the study. Attrititon rate = (# participants who dropped out / total of participants).
Treatment adherence | 7 months
  Finally, number of caps took during the treatment phase will be reported to explore the adherence of treatment.

SECONDARY OUTCOMES:
Probiotics primers | From enrollement to infant 7th day of life
  Evaluate the presence or absence of probiotics in the various samples, i.e. vaginal secretions, meconium and 7-day-old baby's stool, using specific primers to detect strains.

CONTACTS AND LOCATIONS:
Locations (1):
- Centre de recherche du CHUM, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: Yes
Study Protocol, Statistical Analysis Plan (SAP) and informed Consent Form (ICF). No data concerning individual participant will be shared or published.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: The supporting information will be shared before the end of the study.